CLINICAL TRIAL: NCT01991782
Title: The Impact of Telemedicine on Orthopaedic Trauma Patients With Closed Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Manish Sethi, Assistant Professor of Orthopaedics, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120725
Record Dates: First submitted 2012-07-11; First posted 2013-11-25 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Telemedicine; Fracture
Keywords: Telemedicine; Fracture; Orthopaedics
MeSH Terms: conditions — Fractures, Bone | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Control patients with all follow-up visits in person at the Vanderbilt Orthopaedic Trauma clinic (2 weeks, 6 weeks, 3 months, and 6 months post-operative).
- Telemedicine (Experimental): Experimental cohort with two follow-up visits (6 weeks and 6 months) occurring via telemedicine video calls and two follow-up visits (2 weeks and 3 months) occurring in person.
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — Patients in the telemedicine cohort will have two follow-up visits (at 6 weeks and 6 months) through video calls.
  Arms: Telemedicine

SUMMARY:
The purpose of this study is to determine whether telemedicine video calls for follow-up visits between patients and their orthopaedic trauma surgeons has an impact on patient satisfaction, quality of life, and treatment adherence. This study will also assess the feasibility of telemedicine as a medium for follow-up visits.

DETAILED DESCRIPTION:
Patients who are over the age of 18 years with closed fractures treated at Vanderbilt University Medical Center by the Orthopaedic Trauma Department will be recruited into the study into one of two arms: a telemedicine arm in which the patient will have some of his or her visits conducted through video calls, and a control arm in which all of the visits for the patient will be in-person at the Vanderbilt University Orthopaedic Trauma Clinic. Comparisons between the two groups will be made through surveys administered to the patients half-way through the study and at the conclusion of the study, and comparisons will be made using standard statistical tests. The feasibility of telemedicine as a medium for follow-up visits in lieu of in-person visits will be assessed in this study.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years old with closed fracture and having access to telemedicine technology (i.e. high speed Internet) at home

Exclusion Criteria:

* patients as part of vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction and Clinical Outcomes at Conclusion | 6 month
  Surveys will be administered to all patients in both arms of the study at the conclusion of the study to assess patient satisfaction with their treatment arms. Furthermore, all clinical outcomes for patients with be addressed at this point to note fracture healing status, any development of complications, and any redefinition of goals of care.

CONTACTS AND LOCATIONS:
Overall Officials: Manish K Sethi, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States